CLINICAL TRIAL: NCT07321210
Title: Clinical Efficacy and Safety of Radical Nephroureterectomy With Versus Without Template Lymph Node Dissection in High-Risk Upper Tract Urothelial Carcinoma: A Multicenter, Prospective, Randomized Controlled Clinical Trial
Brief Title: Radical Nephroureterectomy With vs Without Template Lymph Node Dissection in High-Risk Upper Tract Urothelial Carcinoma (T-LND UTUC): A Randomized Clinical Trial
Acronym: UTLUND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Second Hospital (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Sun Yat-sen University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Tianjin Third Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TLND-UTUC
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Upper Tract Urothelial Carcinoma; Lymph Node Dissection
Keywords: Upper tract urothelial carcinoma (UTUC); Template Lymph node dissection; Nephroureterectomy; High-risk neoplasm; Randomized Controlled Trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RNU + Template Lymph Node Dissection (Experimental): Participants in this arm will undergo Radical Nephroureterectomy (RNU) combined with template Lymph Node Dissection (LND). The LND will be performed according to a predefined template based on the primary tumor location: renal hilum+para-aortic (left hilar and paraaortic) or renal hilum+para-caval (right hilar, paracaval, and interaortocaval) for renal pelvis/upper ureter; extended to common/external iliac for mid-ureter; and pelvic (common, external, internal iliac, and obturator) for lower ureter. The surgical approach (open, laparoscopic, or robot-assisted) is at the surgeon's discretion.
  Interventions: Procedure: Template Lymph Node Dissection
- RNU + Selective Lymph Node Resection (Active Comparator): Participants in this arm will undergo Radical Nephroureterectomy (RNU) alone. No template lymph node dissection will be performed. However, if intraoperatively identified suspicious and radiographic lymphadenopathy (>1 cm in the short-axis diameter) are present, they may be removed for pathological staging purposes only.
  Interventions: Procedure: Selective Lymph Node Resection

INTERVENTIONS:
Procedure: Template Lymph Node Dissection — A systematic and anatomic-based lymph node dissection performed during radical nephroureterectomy (RNU) for upper tract urothelial carcinoma (UTUC). The dissection boundaries are strictly defined by a pre-specified template according to the primary tumor location: renal hilum+para-aortic (left hilar and paraaortic) or renal hilum+para-caval (right hilar, paracaval, and interaortocaval) for renal pelvis/upper ureter; extended to common/external iliac for mid-ureter; and pelvic (common, external, internal iliac, and obturator) for lower ureter. The goal is potential therapeutic benefit by removing nodal metastatic disease.
  Arms: RNU + Template Lymph Node Dissection
Procedure: Selective Lymph Node Resection — A diagnostic procedure performed during radical nephroureterectomy (RNU). It does not involve a systematic template dissection. The surgeon will only remove intraoperatively identified suspicious and radiographic lymphadenopathy (>1 cm in the short-axis diameter). The primary goal is pathological staging rather than therapeutic clearance of a nodal basin.
  Arms: RNU + Selective Lymph Node Resection

SUMMARY:
The goal of this clinical trial is to learn if adding a template lymph node dissection (TLND) to the standard surgery for upper tract urothelial cancer (UTUC) can improve patient survival and prevent the cancer from recurrence. The main questions it aims to answer are:

Do patients who receive standard surgery with LND live longer without their cancer returning? Is adding LND safe, and how does it affect surgery-related complications? Researchers will compare the group receiving standard surgery plus LND to the group receiving standard surgery alone to see if adding LND is more effective.

Participants will:

Be randomly assigned to one of the two surgical groups. Undergo their assigned surgery and recover in the hospital. Attend regular follow-up visits for checkups and scans for 5 years to monitor for cancer recurrence, with the possibility of long-term follow-up extending to 10 years.

DETAILED DESCRIPTION:
Background： Upper tract urothelial carcinoma (UTUC), encompassing renal pelvic and ureteral carcinomas, is a relatively rare but aggressive malignancy of the urinary system, accounting for 5-10% of all urothelial cancers. Radical nephroureterectomy (RNU) with bladder cuff excision remains the gold standard for treating non-metastatic UTUC. However, prognosis remains poor, particularly for patients with locally advanced disease, due to high rates of recurrence and metastasis. The role of concurrent lymph node dissection (LND) during RNU is one of the most debated topics in UTUC management. While LND is widely accepted in muscle-invasive bladder cancer for its diagnostic and therapeutic benefits, its utility in UTUC lacks high-level evidence. Current guidelines conditionally recommend LND for high-risk UTUC based largely on retrospective data, leading to significant heterogeneity in clinical practice. This multicenter, prospective, randomized controlled trial aims to definitively establish the clinical value of template-based LND in high-risk UTUC.

Objectives：

1. Primary Objectives:

   1. To compare the impact of RNU plus template LND versus RNU alone on disease-free survival (DFS) and overall survival (OS) in patients with high-risk non-metastatic UTUC.
   2. To evaluate and compare the safety profiles of both approaches, including perioperative complications (graded by Clavien-Dindo), operative time, intraoperative blood loss, and length of hospital stay.
2. Secondary Objectives:

   1. To compare non-urothelial tract recurrence-free survival (NU-RFS), intravesical recurrence-free survival (IFS), and cancer-specific survival (CSS) between the two groups.
   2. To establish a lymph node metastasis (pN+) mapping profile for different UTUC tumor locations using template-based LND.
3. Exploratory Objectives:

   1. To identify molecular biomarkers predictive of prognosis using bulk RNA sequencing of prospectively collected tumor tissues.
   2. To develop a lymph node metastasis prediction nomogram based on radiomic data from contrast-enhanced CT, tumor characteristics, lymph node size/location, and clinical symptoms.

Methods：

This is a prospective, multicenter, open-label, randomized controlled trial. A total of 150 eligible patients with high-risk UTUC (cT2-4N0-1M0 or cT1N1M0) will be randomized in a 1:1 ratio to one of two arms:

Experimental Arm (A): RNU + template LND Control Arm (B): RNU + removal of only radiologically or intraoperatively detected lymph nodes >1 cm Stratified randomization will be performed based on tumor location (renal pelvis/upper ureter, mid-ureter, lower ureter) and clinical nodal status (cN0 vs. cN1). Surgical approach (open, laparoscopic, or robotic) will be at the surgeon's discretion, but LND must adhere to predefined anatomical templates.

Patients will be followed for up to 10 years, with regular imaging, urine cytology, and cystoscopy according to a standardized schedule. DFS, OS, and other survival endpoints will be analyzed using Kaplan-Meier methods and Cox proportional hazards models. Safety will be assessed via Clavien-Dindo grading and monitoring of adverse events.

Innovation：

This trial addresses a critical evidence gap in UTUC management by providing the first high-level, prospective, randomized data on the therapeutic efficacy of template LND. Key innovative aspects include:

1. Standardization of LND templates based on tumor location, enhancing surgical consistency and pathological staging.
2. Incorporation of biomarker and radiomic analyses to explore predictive signatures for lymph node involvement and survival.
3. A multicenter design ensuring generalizability and sufficient power to detect clinically meaningful differences in survival outcomes.
4. Potential to establish LND as a standard of care for high-risk UTUC, thereby informing future guidelines and improving oncologic outcomes.

ELIGIBILITY:
Inclusion Criteria:

Signed written informed consent form (ICF). Age > 18 years at the time of ICF signing. Clinical diagnosis of unilateral Upper Tract Urothelial Carcinoma (UTUC) by imaging (enhanced CT or MRI) and/or ureteroscopic biopsy/urinary cytology, and scheduled to undergo Radical Nephroureterectomy (RNU).

Clinical assessment indicating that the tumor and regional lymph nodes are completely resectable, with at least one of the following high-risk features:

1. Locally advanced: Preoperative imaging assessed as cT2 stage or higher (i.e., tumor invades muscularis propria or deeper).
2. High-grade: Preoperative ureteroscopic biopsy pathology confirmed as high-grade urothelial carcinoma (or with squamous differentiation/sarcomatoid differentiation).
3. Moderate or severe hydronephrosis: Ipsilateral moderate or severe hydronephrosis due to tumor obstruction.
4. Large tumor size: Imaging measures maximum tumor diameter > 2 cm.
5. cN1: Imaging suggests regional lymph node short-axis diameter > 1 cm, and the investigator judges it to be resectable.

Presence of at least one measurable lesion according to RECIST v1.1 criteria. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Adequate organ function meeting the following requirements (without use of any blood components or colony-stimulating factors within 14 days):

Bone marrow function: Neutrophils ≥ 1,500/mm³, Platelets ≥ 100,000/mm³, Hemoglobin ≥ 9 g/dL (5.6 mmol/L).

Renal function: Serum creatinine ≤ 1.5 mg/dL and/or Creatinine clearance ≥ 60 mL/min.

Liver function: Total bilirubin ≤ 1.5 × ULN, AST & ALT ≤ 1.5 × ULN. For women of childbearing potential (WOCBP): Must agree to use a highly effective medically approved contraceptive method during the treatment period and for 3 months after treatment ends. A negative serum or urine pregnancy test within 7 days before enrollment is required; must be non-lactating. For non-sterilized male patients: Must agree to use effective contraception with their partner during the treatment period and for 3 months after treatment ends.

Subject voluntarily joins the study, has good compliance, and agrees to undergo safety and survival follow-up.

Exclusion Criteria:

Previous receipt of any anti-tumor therapy for UTUC, including chemotherapy, radiotherapy, immunotherapy, or targeted therapy.

History or concurrent presence of muscle-invasive bladder urothelial carcinoma. Preoperative imaging assesses regional lymph nodes as unresectable: lymph nodes fused into a massive conglomerate, or fully encasing the abdominal aorta/inferior vena cava/pelvic vessels preventing safe separation.

Known bilateral UTUC or hereditary diseases that definitively increase the risk of contralateral upper tract tumors, such as Lynch Syndrome.

Diagnosis of other active malignancies within the past 5 years (except for adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix which have been cured and show no recurrence within 5 years).

Presence of any active autoimmune disease or history of autoimmune disease. Current use of immunosuppressants for immunosuppressive purposes, continued within 2 weeks prior to enrollment.

Poorly controlled cardiac clinical symptoms or diseases. Coagulation abnormalities or bleeding tendency. Presence of specific active gastrointestinal conditions or uncontrolled tumor bleeding.

History of significant bleeding, hemoptysis, or thromboembolic events within specified timeframes.

Active infection or unexplained fever > 38.5°C during screening or before the first dose.

Occurrence of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 4 weeks prior to surgery.

History or current objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severely impaired pulmonary function, etc.

Congenital or acquired immunodeficiency. Participation in another clinical study within 1 month prior to enrollment, or potential receipt of other systemic anti-tumor therapy during the study period.

Known history of psychotropic drug abuse, alcohol abuse, or drug use. Inability or unwillingness to bear the out-of-pocket costs of examinations and treatments. Any other condition deemed by the investigator to make the subject unsuitable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2032-08-30 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | From date of randomization until the date of first documented progression, recurrence, or death from any cause, assessed up to 5 years. (Assessments: every 3 months for the first 2 years, then every 6 months for years 3-5.)
  Time from randomization to the first documented occurrence of disease recurrence (local, regional nodal, or distant metastasis), new urothelial carcinoma in the contralateral upper tract or bladder, or death from any cause, whichever occurs first.
Overall Survival (OS) | From date of randomization until the date of death from any cause, assessed up to 5 years. (Assessments: every 3 months.)
  Time from randomization to death from any cause.
Perioperative Safety | From the date of surgery until 30 days post-operation.
  A composite measure to assess the safety of the surgical procedures, including:
  Incidence and severity of postoperative complications graded by Clavien-Dindo classification.
  Operative time (minutes). Estimated intraoperative blood loss (milliliters). Length of postoperative hospital stay (days).

SECONDARY OUTCOMES:
Non-Urothelial Tract Recurrence-Free Survival (NU-RFS) | From date of randomization until the date of first documented non-urothelial recurrence or death, assessed up to 5 years. (Assessments: every 3 months for the first 2 years, then every 6 months for years 3-5.)
  Time from randomization to the first documented recurrence at a local site, regional lymph nodes, distant metastasis, or death from any cause, whichever occurs first.
Intravesical Recurrence-Free Survival (IFS) | From date of randomization until the date of first documented intravesical recurrence or death, assessed up to 5 years. (Assessments: cystoscopy every 6 months for the first 2 years, then as per protocol.)
  Time from randomization to the first documented occurrence of new urothelial carcinoma in the bladder or contralateral upper tract, or death from any cause, whichever occurs first.
Cancer-Specific Survival (CSS) | Time Frame: From date of randomization until the date of death due to urothelial carcinoma, assessed up to 5 years. (Assessments: every 3 months.)
  Time from randomization to death attributable to urothelial carcinoma.
Lymph Node Metastasis Map | At time of surgery (from final pathological report, approximately 4 weeks post-operation)
  The distribution and positive rate (pN+%) of lymph node metastases, mapped according to the predefined template dissection locations for different primary tumor sites (renal pelvis/upper ureter, mid-ureter, lower ureter).

OTHER OUTCOMES:
Prognostic Biomarker Discovery | Tumor tissue samples are collected at the time of surgery. Biomarker analysis (Bulk RNA-seq) is performed after sample accrual, with the analysis period extending through study completion (up to 10 years).
  Identification of molecular biomarkers predictive of DFS, OS, and CSS through Bulk RNA-sequencing analysis of prospectively collected tumor tissues.
Nomogram for Prediction of Lymph Node Metastasis | Baseline clinical and CT radiomic data are collected preoperatively. Model development and validation are performed after data accrual is sufficient, with the analysis period extending through study completion (up to 10 years).
  Development of a predictive nomogram for lymph node metastasis based on prospectively collected clinical data, CT radiomics features, tumor size/location, and lymph node characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Changyi Quan, MD, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical University Second Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsieh HC, Wang CL, Chen CS, Yang CK, Li JR, Wang SS, Cheng CL, Lin CY, Chiu KY. The prognostic impact of lymph node dissection for clinically node-negative upper urinary tract urothelial carcinoma in patients who are treated with radical nephroureterectomy. PLoS One. 2022 Dec 1;17(12):e0278038. doi: 10.1371/journal.pone.0278038. eCollection 2022. PMID 36454803
- [Background] Bobjer J, Gerdtsson A, Abrahamsson J, Baseckas G, Bergkvist M, Blackberg M, Brandstedt J, Jancke G, Hagberg O, Kollberg P, Lundstrom KJ, Lofgren A, Nyberg M, Rian Martensson L, Saemundsson Y, Stahl E, Sorenby A, Warnolf A, Liedberg F. Location of Retroperitoneal Lymph Node Metastases in Upper Tract Urothelial Carcinoma: Results from a Prospective Lymph Node Mapping Study. Eur Urol Open Sci. 2023 Sep 27;57:37-44. doi: 10.1016/j.euros.2023.09.010. eCollection 2023 Nov. PMID 38020529
- [Background] Li X, Cui M, Gu X, Fang D, Li H, Qin S, Yang K, Zhu T, Li X, Zhou L, Gao XS, Wang D. Pattern and risk factors of local recurrence after nephroureterectomy for upper tract urothelial carcinoma. World J Surg Oncol. 2020 May 30;18(1):114. doi: 10.1186/s12957-020-01877-w. PMID 32473636
- [Background] Zareba P, Rosenzweig B, Winer AG, Coleman JA. Association between lymph node yield and survival among patients undergoing radical nephroureterectomy for urothelial carcinoma of the upper tract. Cancer. 2017 May 15;123(10):1741-1750. doi: 10.1002/cncr.30516. Epub 2017 Feb 2. PMID 28152158
- [Background] Huang J, Qian H, Yuan Y, Cai X, Chen Y, Zhang J, Kong W, Wu X, Cao M, Huang Y, Chen H, Xue W. Prospective Clinical Trial of the Oncologic Outcomes and Safety of Extraperitoneal Laparoscopic Extended Retroperitoneal Lymph Node Dissection at Time of Nephroureterectomy for Upper Tract Urothelial Carcinoma. Front Oncol. 2022 Feb 24;12:791140. doi: 10.3389/fonc.2022.791140. eCollection 2022. PMID 35280720
- [Background] Zhai TS, Jin L, Zhou Z, Liu X, Liu H, Chen W, Lu JY, Yao XD, Feng LM, Ye L. Effect of lymph node dissection on stage-specific survival in patients with upper urinary tract urothelial carcinoma treated with nephroureterectomy. BMC Cancer. 2019 Dec 12;19(1):1207. doi: 10.1186/s12885-019-6364-z. PMID 31830927
- [Background] Messer J, Lin YK, Raman JD. The role of lymphadenectomy for upper tract urothelial carcinoma. Nat Rev Urol. 2011 May 24;8(7):394-401. doi: 10.1038/nrurol.2011.78. PMID 21606972
- [Background] Roscigno M, Brausi M, Heidenreich A, Lotan Y, Margulis V, Shariat SF, Van Poppel H, Zigeuner R. Lymphadenectomy at the time of nephroureterectomy for upper tract urothelial cancer. Eur Urol. 2011 Oct;60(4):776-83. doi: 10.1016/j.eururo.2011.07.009. Epub 2011 Jul 14. PMID 21798659
- [Background] Raza SJ, Miller C, May A, Davaro F, Siddiqui SA, Hamilton Z. Lymph node density for stratification of survival outcomes with node positive upper tract urothelial carcinoma. Can J Urol. 2019 Aug;26(4):9852-9858. PMID 31469641
- [Background] Sato R, Watanabe K, Matsushita Y, Watanabe H, Motoyama D, Ito T, Sugiyama T, Otsuka A, Miyake H. Prognostic assessments in patients with upper tract urothelial carcinoma undergoing radical nephroureterectomy and systematic regional lymph node dissection. Urologia. 2022 Aug;89(3):354-357. doi: 10.1177/03915603211034943. Epub 2021 Jul 29. PMID 34325582
- [Background] Piontkowski AJ, Corsi N, Morisetty S, Majdalany S, Rakic I, Li P, Arora S, Jamil M, Rogers C, Autorino R, Abdollah F. Benefit of lymph node dissection in cN+ patients in the treatment of upper tract urothelial carcinoma: Analysis of NCDB registry. Urol Oncol. 2022 Sep;40(9):409.e9-409.e17. doi: 10.1016/j.urolonc.2022.04.015. Epub 2022 May 24. PMID 35623996
- [Background] Fajkovic H, Cha EK, Jeldres C, Donner G, Chromecki TF, Margulis V, Novara G, Lotan Y, Raman JD, Kassouf W, Seitz C, Bensalah K, Weizer A, Kikuchi E, Roscigno M, Remzi M, Matsumoto K, Breinl E, Pycha A, Ficarra V, Montorsi F, Karakiewicz PI, Scherr DS, Shariat SF. Prognostic value of extranodal extension and other lymph node parameters in patients with upper tract urothelial carcinoma. J Urol. 2012 Mar;187(3):845-51. doi: 10.1016/j.juro.2011.10.158. Epub 2012 Jan 15. PMID 22248522
- [Background] Siegel RL, Kratzer TB, Giaquinto AN, Sung H, Jemal A. Cancer statistics, 2025. CA Cancer J Clin. 2025 Jan-Feb;75(1):10-45. doi: 10.3322/caac.21871. Epub 2025 Jan 16. PMID 39817679
- [Background] Cui Y, Lu Y, Wu J, Quan C. Benefits of lymphadenectomy for upper tract urothelial carcinoma only located in the lower ureter: a bicentre retrospective cohort study. Front Oncol. 2023 Apr 14;13:1115830. doi: 10.3389/fonc.2023.1115830. eCollection 2023. PMID 37124512
- [Background] Lee HY, Chang CH, Huang CP, Yu CC, Lo CW, Chung SD, Wu WC, Chen IA, Lin JT, Jiang YH, Lee YK, Hsueh TY, Chiu AW, Chen YT, Lin CM, Tsai YC, Chen WC, Chiang BJ, Huang HC, Chen CH, Huang CY, Wu CC, Lin WY, Tseng JS, Ke HL, Yeh HC. Is Lymph Node Dissection Necessary During Radical Nephroureterectomy for Clinically Node-Negative Upper Tract Urothelial Carcinoma? A Multi-Institutional Study. Front Oncol. 2022 Apr 29;12:791620. doi: 10.3389/fonc.2022.791620. eCollection 2022. PMID 35574295
- [Background] Xia HR, Li SG, Zhai XQ, Liu M, Guo XX, Wang JY. The Value of Lymph Node Dissection in Patients With Node-Positive Upper Urinary Tract Urothelial Cancer: A Retrospective Cohort Study. Front Oncol. 2022 Jun 16;12:889144. doi: 10.3389/fonc.2022.889144. eCollection 2022. PMID 35785156
- [Background] Dlubak A, Karwacki J, Logon K, Tomecka P, Brawanska K, Krajewski W, Szydelko T, Malkiewicz B. Lymph Node Dissection in Upper Tract Urothelial Carcinoma: Current Status and Future Perspectives. Curr Oncol Rep. 2023 Nov;25(11):1327-1344. doi: 10.1007/s11912-023-01460-y. Epub 2023 Oct 6. PMID 37801187
- [Background] Li Q, Wei P, Kang Y, Li X, Zhang H, Yang J, Sun J. To explore the risk factors of lymphovascular invasion in patients with upper tract urothelial carcinoma and construct a prediction model. Front Oncol. 2025 Mar 25;15:1568774. doi: 10.3389/fonc.2025.1568774. eCollection 2025. PMID 40201351
- [Background] Seisen T, Shariat SF, Cussenot O, Peyronnet B, Renard-Penna R, Colin P, Roupret M. Contemporary role of lymph node dissection at the time of radical nephroureterectomy for upper tract urothelial carcinoma. World J Urol. 2017 Apr;35(4):535-548. doi: 10.1007/s00345-016-1764-z. Epub 2016 Jan 25. PMID 26809456
- [Background] Inokuchi J, Kuroiwa K, Kakehi Y, Sugimoto M, Tanigawa T, Fujimoto H, Gotoh M, Masumori N, Ogawa O, Eto M, Ohyama C, Yamaguchi A, Matsuyama H, Ichikawa T, Asano T, Mizusawa J, Eba J, Naito S. Role of lymph node dissection during radical nephroureterectomy for upper urinary tract urothelial cancer: multi-institutional large retrospective study JCOG1110A. World J Urol. 2017 Nov;35(11):1737-1744. doi: 10.1007/s00345-017-2049-x. Epub 2017 May 15. PMID 28508102
- [Background] Dominguez-Escrig JL, Peyronnet B, Seisen T, Bruins HM, Yuan CY, Babjuk M, Bohle A, Burger M, Comperat EM, Gontero P, Lam T, MacLennan S, Mostafid H, Palou J, van Rhijn BWG, Sylvester RJ, Zigeuner R, Shariat SF, Roupret M. Potential Benefit of Lymph Node Dissection During Radical Nephroureterectomy for Upper Tract Urothelial Carcinoma: A Systematic Review by the European Association of Urology Guidelines Panel on Non-muscle-invasive Bladder Cancer. Eur Urol Focus. 2019 Mar;5(2):224-241. doi: 10.1016/j.euf.2017.09.015. Epub 2017 Nov 20. PMID 29158169
- [Background] Yanagisawa T, Kawada T, von Deimling M, Laukhtina E, Kimura T, Shariat SF. Need for and extent of lymph node dissection for upper tract urothelial carcinoma: an updated review in 2023. Curr Opin Urol. 2023 Jul 1;33(4):258-268. doi: 10.1097/MOU.0000000000001097. Epub 2023 Apr 3. PMID 37014743
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Soukup V, Capoun O, Cohen D, Hernandez V, Babjuk M, Burger M, Comperat E, Gontero P, Lam T, MacLennan S, Mostafid AH, Palou J, van Rhijn BWG, Roupret M, Shariat SF, Sylvester R, Yuan Y, Zigeuner R. Prognostic Performance and Reproducibility of the 1973 and 2004/2016 World Health Organization Grading Classification Systems in Non-muscle-invasive Bladder Cancer: A European Association of Urology Non-muscle Invasive Bladder Cancer Guidelines Panel Systematic Review. Eur Urol. 2017 Nov;72(5):801-813. doi: 10.1016/j.eururo.2017.04.015. Epub 2017 Apr 28. PMID 28457661
- [Background] Kondo T, Hara I, Takagi T, Kodama Y, Hashimoto Y, Kobayashi H, Iizuka J, Omae K, Yoshida K, Tanabe K. Template-based lymphadenectomy in urothelial carcinoma of the renal pelvis: a prospective study. Int J Urol. 2014 May;21(5):453-9. doi: 10.1111/iju.12417. PMID 24754341
- [Background] Matin SF, Sfakianos JP, Espiritu PN, Coleman JA, Spiess PE. Patterns of Lymphatic Metastases in Upper Tract Urothelial Carcinoma and Proposed Dissection Templates. J Urol. 2015 Dec;194(6):1567-74. doi: 10.1016/j.juro.2015.06.077. Epub 2015 Jun 19. PMID 26094807
- [Background] Masson-Lecomte A, Birtle A, Pradere B, Capoun O, Comperat E, Dominguez-Escrig JL, Liedberg F, Makaroff L, Mariappan P, Moschini M, Rai BP, van Rhijn BWG, Shariat SF, Smith EJ, Teoh JYC, Soukup V, Wood R, Xylinas EN, Soria F, Seisen T, Gontero P. European Association of Urology Guidelines on Upper Urinary Tract Urothelial Carcinoma: Summary of the 2025 Update. Eur Urol. 2025 Jun;87(6):697-716. doi: 10.1016/j.eururo.2025.02.023. Epub 2025 Mar 20. PMID 40118741

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT07321210/Prot_SAP_000.pdf
  • Informed Consent Form (2025-08-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT07321210/ICF_001.pdf